CLINICAL TRIAL: NCT01233817
Title: Pilot Study of Progressive Strength Training in Spinal Muscular Atrophy
Brief Title: Progressive Strength Training in Spinal Muscular Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39995
Record Dates: First submitted 2010-10-19; First posted 2010-11-03 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Muscular Atrophy, Spinal
Keywords: Spinal muscular atrophy; Neuromuscular disorder; Progressive strength training; Children
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spinal muscular atrophy (Experimental): Children and adolescents with diagnosis of SMA type II or III. The intervention group (the only arm/group in this pilot study) receives a home-based, supervised, 12-week progressive strength-training program.
  Interventions: Other: Progressive strength training

INTERVENTIONS:
Other: Progressive strength training — the systematic increase in resistance weights

SUMMARY:
The proposed feasibility study is necessary to test if children and young adults will participate in and adhere to a 12-week, home-based, supervised progressive strength training exercise program and to obtain preliminary data that will subsequently allow us to determine the safety and impact of strength training in spinal muscular atrophy. Our pilot study will address 3 aims: (1) Ascertain the feasibility of, and potential barriers to, participation in and adherence to a 12-week home-based, supervised, progressive strength training exercise program in children and young adults aged 5-21 years with SMA types II and III; (2) Determine the safety and tolerability of progressive strength training in a pilot study sample of children and young adults with SMA types II and III; and (3) Determine candidate outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* age 5-21 years
* diagnosis of SMA type II or III
* at least antigravity strength in elbow flexors
* ability to follow commands and stay on task
* place of residence within a 60-minute or 60-mile drive of the University of Utah

Exclusion Criteria:

* planned surgery or out-of-town trips during the proposed intervention period
* inability to travel to study center for testing
* neurological diagnosis other than SMA

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aga Lewelt, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2010 until February 2012. Some participants were recruited during clinic visits and others contacted us after being informed of the study
Pre-assignment Details: This was a pilot study and all participants were in the treatment group
Groups:
- Spinal Muscular Atrophy: Children and adolescents with diagnosis of SMA type II or III
Period: Overall Study
Arm/Group | Spinal Muscular Atrophy
Started | 12
Completed | 9
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Muscular Atrophy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.56 (3.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Strength
Description: Primary Outcome Measure was muscle strength. Strength was measured using a fixed myometry evaluation, quantitative muscle analysis (QMA). QMA utilizes a relative fixed point for the participant to exert effort. Each muscle of interest was tested using QMA.
Time Frame: 12 weeks
Measure: Median (95% Confidence Interval); unit: kilograms
Arm/Group | Spinal Muscular Atrophy
Number analyzed (Participants) | 9
kilograms | 0.39 [-0.5 to 1.1]

ADVERSE EVENTS:
Arm/Group | Spinal Muscular Atrophy
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
This was a pilot study with only one arm, the treatment arm. This is an inherent limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes